CLINICAL TRIAL: NCT02407561
Title: Prospective Validation Study Under CLIA-compliant SOPs for the Proprietary Rectal and Anal Cancer Protein Expression Assays
Brief Title: Prospective Validation Study for the Proprietary Rectal and Anal Cancer Protein Expression Assays
Status: Terminated | Type: Observational
Why Stopped: Futility - unable to secure sites and samples for participation
Sponsor: Castle Biosciences Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: Protocol_CBI_RC_PVS
Record Dates: First submitted 2015-03-26; First posted 2015-04-03 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2016-07

CONDITIONS: Rectal Adenocarcinoma; Anal Adenocarcinoma; Anal Squamous Cell Carcinoma
Keywords: rectal; adenocarcinoma; DecisionDx
MeSH Terms: conditions — Rectal Neoplasms; Anus Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Formalin Fixed Paraffin Embedded (FFPE) H&E stained tumor samples(biopsy and resection) cDNA- tumor sample IHC Stained FFPE- tumor samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with locally advanced rectal and esophageal carcinomas typically undergo neoadjuvant chemoradiation therapy prior to surgical resection. While response rates to this treatment differ among these three cancers, generally 20-25% of patients exhibit minimal or no response to preoperative chemoradiation therapy while 20-30% exhibit a complete pathologic response, and the remainder receiving a partial response.

This will be a multi-center study of patients with newly diagnosed rectal adenocarcinoma, or anal squamous cell carcinoma (SCC) who will undergo neoadjuvant chemoradiation prior to surgery. The tumor from these patients will be tested to determine whether response to neoadjuvant chemoradiation can be accurately predicted.

DETAILED DESCRIPTION:
Patients with locally advanced rectal and esophageal carcinomas typically undergo neoadjuvant chemoradiation therapy prior to surgical resection, although the specific chemoradiation regimens may vary. While response rates differ among these three cancers, generally 20-25% of patients exhibit minimal or no response to preoperative chemoradiation therapy while 20-30% exhibit a complete pathologic response, and the remainder receiving a partial response.

In esophageal adenocarcinoma, patients who achieve a complete response tend to have a significantly longer overall survival than those who do not achieve a complete response. Similar data exists for rectal cancer that the degree of responsiveness to chemoradiation regimens dictates survival outcome in patients.

If patients with distinct response profiles can be identified before treatment starts, personalized regimens can be delivered to maximize the benefit in each patient population: complete responders may be spared post-treatment surgical resection, while non responders may consider avoiding ineffective chemoradiation prior to surgery.

Target Population:

Subjects with newly diagnosed rectal adenocarcinoma, or anal squamous cell carcinoma (SCC) who will undergo neoadjuvant chemoradiation prior to surgery.

350 patient samples will be included in this validation study, given the predicted 25% population size that exhibit pathologic complete response (pathCR) to pre-operative chemo/radiation therapy, and the predicted 25% population size that have no response (exCTRT) to pre-operative treatment.

Study Design:

This will be a multi-center prospective study of up to 350 patients, each having both pre-treatment (prior to chemoradiation) unstained sections on charged slides from the FFPE block that was used for diagnosis of rectal or anal cancer and sections of unstained, post-surgical, resected tissue (pathologic confirmation of treatment response based upon endoscopy or ultrasound can be accepted in place of post-surgical resected tissue). Per the CLIA-compliant SOPs (Appendix A), one slide will be stained with H&E to define the area of tumor within the tissue, and the remaining slides will be used for immunohistochemical (IHC) detection of the biomarkers described above to assess the performance of the proprietary IHC assay. Any remaining slides not used for IHC staining will be used for a parallel gene expression discovery effort using TaqMan high throughput RT-PCR analysis (Appendix B, Sub-study 1).

The proprietary assay will be performed under CLIA certified standard operating procedures. The individual assay results, treatment effect, actual survival data, and other clinical data will be analyzed. Initial labeling index data will be used to develop a training set and unique algorithmic approach specifically applicable to rectal and anal carcinoma. The remaining samples will be embargoed for use as an independent test set.

Associated clinical data will be collected :

1. Age of patient at diagnosis
2. Gender
3. Date of diagnosis rectal/anal cancer
4. Histotype of rectal/anal cancer
5. Stage of rectal/anal cancer at diagnosis and again after neoadjuvant treatment (if available)
6. Details of imaging performed
7. Clinical and histopathalogical features of primary tumor
8. Details of any genetic testing performed.
9. Extent/approach of surgical resection
10. Date of last contact
11. First progression documentation (Y/N). If yes, location of first progression and date of first progression.
12. Method of diagnosis of first progression.
13. Death documentation (Y/N). If yes, date of death, cause of death.
14. Pre-operative treatments received:

    1. Start/stop date of radiation
    2. Radiation dose, fractions given, interruptions to treatment (Y/N), reasons if Yes
    3. Start/stop date of chemotherapy
    4. Chemotherapeutic agent(s) and doses, interruptions to treatment (Y/N), reasons if Yes
15. Post-surgical treatments received:

    1. Start/stop date of radiation
    2. Radiation dose, fractions given, interruptions to treatment (Y/N), reasons if Yes
    3. Start/stop date of chemotherapy
    4. Chemotherapeutic agent(s) and doses, interruptions to treatment (Y/N), reasons if Yes

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically confirmed stage II and III rectal adenocarcinoma or subjects with histologically confirmed stage II and III anal SCC
2. Subjects greater than 18 years of age.
3. Subjects who will undergo prescribed neoadjuvant chemotherapy and/or radiotherapy and have surgical resection prior to further treatment or pathologic confirmation of treatment response using endoscopy or ultrasound.
4. Subjects with:

   * twenty (20) unstained sections on charged slides available from tumor block (FFPE) used for the diagnosis of rectal/anal carcinoma or adjacent to this block (pre-neoadjuvant biopsy sample); and
   * four (4) unstained slides available from post-chemoradiation surgery to allow for blinded pathology review and assessment of pathCR, partial CR, or exCTRT. Slides from surgical resection are not necessary in cases with documented post-surgical determination of response by ultrasound or endoscopy.
5. Subjects willing to complete study follow up for outcomes.
6. Subjects from who informed consent can be obtained.

Exclusion Criteria:

1. Subjects with carcinoma in situ or Stage I rectal/anal carcinoma.
2. Subjects with Stage IV rectal/anal carcinoma.
3. Subjects with diagnosis of other malignant tumors with the exception of non-melanoma skin cancers cured by resection only.
4. Subjects that have received prior chest or upper abdomen radiotherapy and/or system chemotherapy within the past 5 years
5. Subjects who are unwilling to complete study follow up
6. Employees and family members of Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with newly diagnosed rectal adenocarcinoma, or anal squamous cell carcinoma (SCC) who will undergo neoadjuvant chemoradiation prior to surgery.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2015-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Validate the proprietary rectal and anal carcinoma immunohistochemistry protocols under CLIA compliant SOPs, in order to predict response to pre-operative chemoradiation treatment for patients with rectal/ anal carcinoma. | at time of surgical resection (visit 3) - review of resected tumor
  Post treatment tissue will be reviewed by independent pathologist for Treatment Response grade.
Gene expression profiling will be undertaken to determine if RNA is a superior biomarker to protein | at time of enrollment (visit 1) tissue will be sent for testing
  once testing done the results will be compared to the resection Treatment Response grade determined by pathologist.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cook, PhD, Principal Investigator — Castle Biosciences Inc.
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States